CLINICAL TRIAL: NCT06666179
Title: A Phase 1, Placebo-controlled, Randomized, Observer-blind Study to Describe the Safety, Reactogenicity and Immunogenicity of a Bivalent Recombinant RSV Vaccine (SCB-1019T) in Children 2 to <6 Years of Age
Brief Title: Safety and Immunogenicity Study of SCB-1019T in Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated during the EC submission process prior to the enrolment
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-1019-003
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: RSV Infection
Keywords: RSV vaccine
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (low dose SCB-1019T ) (Experimental): 24 children (2-<6 years of age) will receive low-dose unadjuvanted SCB-1019T at Day 1
  Interventions: Biological: low dose SCB-1019T
- Group 2 (adjuvanted low dose SCB-1019T) (Experimental): 24 children (2-<6 years of age) will receive low-dose adjuvanted SCB-1019T at Day 1
  Interventions: Biological: adjuvanted low dose SCB-1019T
- Group 3 (Placebo) (Placebo Comparator): 8 children (2-<6 years of age) will receive placebo at Day 1
  Interventions: Other: Placebo
- Group 4 (high dose SCB-1019T) (Experimental): 24 children (2-<6 years of age) will receive high-dose unadjuvanted SCB-1019T at Day 1
  Interventions: Biological: high dose SCB-1019T
- Group 5 ( adjuvanted high dose SCB-1019T) (Experimental): 24 children (2-<6 years of age) will receive high-dose adjuvanted SCB-1019T at Day 1
  Interventions: Biological: adjuvanted high dose SCB-1019T
- Group 6 (Placebo) (Placebo Comparator): 8 children (2-<6 years of age) will receive placebo at Day 1
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: low dose SCB-1019T — Bivalent Recombinant Respiratory Syncytial Virus (RSV) Vaccine (CHO Cell) (SCB-1019T)
  Arms: Group 1 (low dose SCB-1019T )
Biological: adjuvanted low dose SCB-1019T — Bivalent Recombinant Respiratory Syncytial Virus (RSV) Vaccine (CHO Cell) (SCB-1019T)
  Arms: Group 2 (adjuvanted low dose SCB-1019T)
Biological: high dose SCB-1019T — Bivalent Recombinant Respiratory Syncytial Virus (RSV) Vaccine (CHO Cell) (SCB-1019T)
  Arms: Group 4 (high dose SCB-1019T)
Biological: adjuvanted high dose SCB-1019T — Bivalent Recombinant Respiratory Syncytial Virus (RSV) Vaccine (CHO Cell) (SCB-1019T)
  Arms: Group 5 ( adjuvanted high dose SCB-1019T)
Other: Placebo — 0.9% NaCl saline placebo
  Arms: Group 3 (Placebo); Group 6 (Placebo)

SUMMARY:
This phase 1 study in Australia will evaluate the safety, reactogenicity and immunogenicity of the Bivalent Recombinant Respiratory Syncytial Virus (RSV) Vaccine (CHO Cell) (SCB-1019T) in children 2-<6 years of age.

DETAILED DESCRIPTION:
This Phase 1 randomized, placebo-controlled, observer-blind study will evaluate the safety, reactogenicity and immunogenicity of different formulations of SCB-1019T vaccine in children 2-<6 years of age. A placebo is used as a control in the study because there is no licensed RSV comparator vaccine available for young children globally.

ELIGIBILITY:
Inclusion Criteria:

• Male and female participants 2 to <6 years of age at Visit 1. • Parents/guardians of participants willing and able to provide written informed consent and comply with study requirements, including all scheduled visits, vaccination, laboratory tests, and other study procedures. • Healthy participants as determined by medical history, physical examination, and clinical judgment of the investigator.

For full inclusion criteria, please refer to full protocol.

Exclusion Criteria:

* Acute disease or fever (≥38°C) at time of vaccination. For participants with minor illness and/or fever at the time of vaccination, Visit 1 may be rescheduled.
* Evidence of chronic diseases including hepatitis, bleeding disorders, metabolic diseases, autoimmune diseases, neurological conditions that impair respiratory functions, genetic disorders that increase the risk of severe respiratory diseases, major congenital malformations, cardiac and lung diseases or reactive airway diseases.

For full Exclusion criteria, please refer to full protocol

Ages: 24 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate porportion of participants with solicied AEs of SCB-1019T vaccine | Within 7 days after vaccination
  Porportion of participants with local and systemic solicied AEs
Evaluate porportions of participants with unsolicited AEs of SCB-1019T vaccine | Within 28 days after vaccination
  Porportions of participants with unsolicited AEs
Evaluate porportions of participants with SAEs, AESIs, MAAEs, AEs leading to early termination from the study of SCB-1019T vaccine | Throughout the study period, from enrollment to 6 months follow up
  Porportions of participants with SAEs, AESIs, MAAEs, AEs leading to early termination from the study

CONTACTS AND LOCATIONS:
Locations (1):
- The Kids Research Institute, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided